CLINICAL TRIAL: NCT03409302
Title: The Effectiveness of a Brief Digital ACT Intervention for Chronic Pain
Brief Title: Internet-based Acceptance and Commitment Therapy for Chronic Pain
Acronym: ALGEApp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Maria Karekla, Licensed Clinical Psychologist, Assistant Professor, Peer reviewed ACT trainer, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K3_K1_0c
Record Dates: First submitted 2017-04-06; First posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Chronic Pain
Keywords: ACT; digital intervention; web-based; adherence
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind (subject, outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ALGEapp (Brief i-ACT intervention) (Experimental): The intervention builds on a previously unpublished face-to-face protocol for greek-speaking chronic pain sufferers (developed by Karekla & Vasiliou, 2013) and has been simplified and modified to produce a self-help digital internet-based modality, namely the ALGEApp. ALGEApp consists of a total of 4 approximately one-hour sessions, which are structured to be completed by the users in sequence within a time frame of 2-8 weeks (depending on the rate of completion by each user). The intervention is guided, which implies that an animated character (an Avatar) guides the user throughout the whole duration of the intervention. ALGEApp contains experiential and audiovisual psycho-educational material based on ACT, adopted for the Greek-Cypriot culture.
  Interventions: Behavioral: ALGEApp (Brief iACT intervention)
- Active Control group (Active Comparator): The Active control group will have access only to limited component of the ALGEApp intervention, namely the Bonus section, which contains limited psycho-educational information regarding pain management.
  Interventions: Behavioral: Active control group

INTERVENTIONS:
Behavioral: ALGEApp (Brief iACT intervention) — Participants will be randomly assigned to one of the two groups: brief i-ACT intervention or active control group. The i-ACT intervention participants will be encouraged to login the website platform with their credentials and to complete 4 weekly sessions (1 session per week) which lasts about 1 hour each. Participants will be guided by a 3D- animated Avatar who adopts the role of a facilitator.
  Other Names: ALGEApp
  Arms: The ALGEapp (Brief i-ACT intervention)
Behavioral: Active control group — Participants will be randomly assigned to one of the two groups: brief i-ACT intervention or active control group. The active control group will have access, through the same platform. only to limited online psycho-educational information regarding pain. Active control group will complete pre-treatment and post-treatment questionnaires in parallel with the intervention group.
  Arms: Active Control group

SUMMARY:
Acceptance and Commitment Therapy (ACT) delivered face-to-face is an empirically supported intervention for the management of chronic pain (CP). However, increasing demands for cost reduction in healthcare services in addition to obstacles regarding physical access to treatment, highlight the need for innovative, cost-reducing, digital self-management interventions. Poor user engagement nonetheless, is a significant challenge often faced in digital interventions, which often results in poor adherence or even non-completion in treatment. In addition, very few digital trials appear to plan for adherence a-priori, when designing an intervention. To date there are only two ACT-based digital interventions for CP demonstrating significant improvements in pain-related disability and increased functioning, yet with small to medium effect sizes and poor adherence rates. However, several limitations of the studies such as the absence of a-priori adherence planning and lack of investigation of underlying mechanisms, makes it difficult to draw clear conclusions on the effectiveness of this new treatment modality for chronic pain and warrants further research. This study seeks to: a) explore how a brief adherence-planned digital ACT-based intervention for CP management, compared to an active control group and a wait-list control group improves targeted study outcomes such as functioning and quality of life, and b) investigate which processes of change mediate the targeted study outcomes. It is hypothesized that the brief ACT-based digital intervention in comparison to the active control group and wait-list will result in increased functioning, improved quality of life and reduced pain intensity. The results of the study are expected to shed more light on the utility of planning for adherence in digital interventions and effectiveness of ACT-based digital interventions and their underlying mechanisms in the management of CP.

DETAILED DESCRIPTION:
A growing body of evidence demonstrates that clinic-based interventions can be effectively used to treat pain-related interference in the daily life of chronic pain sufferers. Acceptance and Commitment Therapy (ACT) delivered face-to-face is an empirically supported intervention for the management of chronic pain (CP). The increasing demands for cost reduction for services in the healthcare system and obstacles regarding physical access to treatment highlight the need for innovative, cost-reducing, self-management interventions. In addition, the idea of home-based self-management support seems appealing to a significant number of sufferers of chronic conditions such as chronic pain. Digital interventions might present with feasible means to overcome many barriers such as physical access to treatment or financial obstacles while helping improve health care for persons with chronic pain in the convenience of their space and time.

A considerable number of studies have demonstrated the effectiveness of psychological digitalised interventions (the majority cognitive and behavioural based) in improving chronic pain management, reducing pain intensity, catastrophizing and improving functioning. However, support for the effectiveness of digital interventions is tempered by a plethora of evaluations that report users often fail to adhere to online interventions. Almost twice as many users appear to dropout from internet-based interventions compared to the traditional face-to-face interventions suggesting that users become disengaged and unmotivated early on in these interventions. A-priori planning for maximised user engagement and consequently adherence, using a theoretical framework such as persuasive technology, is desirable in digital interventions that aim to combat the problem of low adherence.

To date, there are only two studies that have examined the effectiveness of ACT-based digital interventions (iACT) for chronic pain management, demonstrating significant improvements in pain-related disability and increased functioning. Despite these encouraging findings, to our knowledge, no iACT study has appropriately addressed the problem of low adherence, which has resulted in low adherence and high attrition rates in both of the ACT trials. Also, none of the two studies has investigated the impact of adherence on treatment outcomes or investigated the underlying ACT mechanisms of change on treatment outcomes within a digital tested framework. Furthermore, there have been very few attempts to examine the effectiveness of brief (< 6 sessions) interventions in the field of ACT and CP, yet none exists in the field of iACT and CP.

The present study seeks to: a) design an innovative Avatar-led digitalised brief intervention based on a culturally sensitive ACT face-to-face protocol developed in a previous project, b) recruit and offer online treatment to community-based chronic pain sufferers, c) explore how a brief iACT intervention for CP management, compared to a waitlist control group (medical treatment as usual) and an active control group (limited access to pain-related psycho-educational information) improves targeted study outcomes (e.g., functioning and quality of life etc.), d) investigate which processes of change mediate the targeted study outcomes and e) investigate the relationship between adherence to the intervention and treatment outcomes. Assessments of chronic pain users' daily functioning (primary outcome), quality of life, affective components, pain intensity (secondary outcomes), therapeutic process measures (e.g., psychological flexibility, acceptance, defusion), will be assessed before and following treatment completion, and after 3, 6 and 12 months. In addition, user satisfaction and web-metrics (number of logins/modules/activities completed, time spent online etc.) will be assessed to examine the relationship between adherence and treatment outcomes.

It is hypothesised that the brief iACT in comparison with the two control groups will result in increased functioning, improved quality of life and reduced pain intensity mediated by the mechanisms of change of psychological flexibility, acceptance and defusion. In addition, it is hypothesized that users with increased adherence will result in significantly improved treatment outcomes as compared to users with poor adherence. The results of this study are expected to revolutionize the implementation and treatment effectiveness of brief iACT interventions in the field of chronic pain management. Furthermore, the investigators attempt to contribute to the literature concerning the improvement of designing and planning for digital interventions that target improved user engagement and adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. At least 3 months chronic pain duration,
3. At least a pain intensity score of ≥ 4 prior to the intervention (assessed by an 11 point numeric rating scale (NRS; Dworkin et al., 2005) ranging from (0) 'no pain' to (10) 'pain as bad as the participant can imagine'.
4. Users to have undergone medical assessment within one year,
5. Official medical diagnosis on the type of chronic pain that users suffer from,
6. Regular access to a computer/tablet and internet
7. Sufficient knowledge of the Greek language.

Exclusion Criteria:

1. Comorbidity with a serious medical condition other than chronic non-malignant pain (e.g., complete paraplegia or tetraplegia, heart or vascular diseases, malignant pain such as cancer etc.), which may interfere with participation. A neurologist will be consulted and candidates will be excluded if their medical condition is regarded as significantly interfering with their participation.
2. Recent episodes of active psychosis, manic episodes, substance use disorder and suicidal ideation. Assessment will take place using selected single items from mini-SCID (mini - Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders Karekla & Panayiotou 2010). Candidates who respond positively to one or more of the assessed mini-SCID items will be excluded from further participation and will receive information over the phone with advice to seek help, along with relevant information on available services from their local community mental health services or their general practitioner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Changes in daily functioning assessed with the Greek Brief Pain Inventory: Interference sub-scale (G-BPI; Mystakidou, Mendoza, Tsilika, Befon, Parpa et al., 2001; Original: Cleeland & Ryan; 1994) | Change in levels of daily functioning from baseline through study completion (approximately 2 months) and at 6 and 12 months post completion. Data will be reported for study completion (approximately 2 months), 6 months and 12 months
  This is a subscale of the Greek-Brief Pain Inventory which is a pain assessment tool developed to assess pain severity and interference which has been previously translated and validated in a Greek chronic pain sample. Pain severity is of secondary focus within the study and will be assessed by a numerical rating scale as described later. The interference subscale will only be used to assess how pain interferes in several areas of daily functioning of chronic pain sufferers. It contains 7-items rated on a Likert-type scale from 0="does not interfere" to 10="completely interferes". The G-BPI presents with good internal consistency (α=.85 for interference) and sufficient validity with theoretically-consistent instruments.

SECONDARY OUTCOMES:
Changes in the quality of life assessed by the World Health Organisation Quality of Life-BREF Questionnaire (WHOQOL-BREF; The WHOQOL Group, 1998) | Change in levels of quality of life from baseline through study completion (approximately 2 months) and at 6 and 12 months post completion. Data will be reported for study completion (approximately 2 months), 6 months and 12 months
  The WHOQOL assesses an individual's quality of life (QoL). The instrument is a self-report 26-item inventory of generic QoL and is divided into four subscales: physical health, mental health, social relationships, and social environment. Higher scores indicate better QoL. WHOQOL-BREF has been previously translated and validated in Greek (Ginieri-Coccossis, Triantafillou, Tomaras, Soldatos, Mavreas, & Christodoulou, 2012) with satisfactory internal consistency between the domains ranging from (Cronbach's α=.66 - .80) and overall QoL (α= .87) and seems to function well for assessing QoL in clinical and general populations.
Changes in the levels of psychological distress assessed by the Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983) | Change in levels of depression and anxiety symptoms from baseline through study completion (approximately 2 months) and at 6 and 12 months post completion. Data will be reported for study completion (approximately 2 months), 6 months and 12 months
  HADS is a 14-item questionnaire assessing levels of depression and anxiety symptomatology, considered unbiased by coexisting medical conditions (Snaith, 1987). Each subscale consists of 7 items rated on a 4-point scale (0-3). Higher scores indicate greater anxiety and depression. The Greek version presents with high internal consistency (α=.88) and validity (Michopoulos, et al., 2008).

OTHER OUTCOMES:
Changes in avoidance of pain levels as assessed by the Greek Psychological Inflexibility in Pain Scale (G-PIPS-II; Vasiliou et al., under submission; Original: Wicksell et al., 2010) | Change in levels of psychological flexibility from baseline through study completion (approximately 2 months) and at 6 and 12 months post completion. Data will be reported for study completion (approximately 2 months), 6 months and 12 months
  G-PIPS-II contains 12 items assessing psychological inflexibility and is comprised of two subscales: a) avoidance of pain (8 items), examines behaviors that lead to avoidance of pain and related distress; and b) cognitive fusion (4 items), assesses how CP sufferers' thoughts about an event can lead to avoidance of pain or distress. Items are rated on a 7-point Likert-type scale, with 1="never true" and 7="always true". The scale demonstrates good psychometric properties (Wicksell et al., 2010) and high internal consistency (α = .88) and validity with associated constructs in its Greek version.
Changes in the levels of pain acceptance as assessed via the Greek Chronic Pain Acceptance Questionnaire (G-CPAQ; Vasiliou et al., under review; Original: McCracken et al., 2004) | Change in levels of pain acceptance from baseline through study completion (approximately 2 months) and at 6 and 12 months post completion. Data will be reported for study completion (approximately 2 months), 6 months and 12 months
  assesses pain acceptance in two sub-factors: activity engagement (4 items) and pain willingness (4 items). Activity engagement, examines the degree to which participants engage in meaningful activity even in the presence of pain. Pain willingness, assesses the degree to which individuals allow pain to occur without trying to change, control, or struggle with it. The G-CPAQ is rated on a 7-point Likert scale (0=never true to 6=always true) and yields a total sum with a range of 0-48. Higher total score suggests greater pain acceptance, whereas higher subscale scores denote greater activity engagement and pain willingness (McCracken et al., 2014). The G-CPAQ presents with high reliability (Cronbach's a=.80) and sufficient construct validity with theoretically-related constructs.
Changes in the levels of defusion with pain-related thoughts as assessed via Cognitive Defusion Stamp (Karekla & Nicolaou, 2011) | Change in levels of defusion at 4 points from baseline through completion (approximately once every week, prior to each session). Data will be reported once when study is completed (approximately 2 months after baseline)
  ): This is a figurative measure developed and used previously in several studies (e.g., Savvide & Karekla, 2015) to assess weekly changes in participants' cognitive defusion related to sabotaging thoughts. It was found to be sensitive to session-to-session changes and correlated significantly with other cognitive defusion measures. In this study the Cognitive Defusion Stamp will be used to assess how fused participants are with thoughts related to pain. CP sufferers will use a circular electronic stamp to show where they consider themselves to be in relation to an existing stamp, which represents pain related thoughts (i.e. "How fused is the participant today with their pain related thoughts?"). The mean distance in mm between the centers of the 2 circles are measured. The longer the distance between the two centers the more defusion from thoughts.
Changes in the levels of satisfaction with treatment as assessed by the Greek Client Satisfaction Questionnaire (CSQ-8; Flora & Stalikas; 2012; Larsen, Attkinson, Hargreaves & Nguyen, 1979) | Change in levels of satisfaction from baseline through study completion (approximately 2 months). Data will be reported once when study is completed (approximately 2 months after baseline)
  G-CSQ-8 will be used to assess participants' evaluation of the intervention and satisfaction. The scale demonstrated high internal consistency (α= .83). Items are rated on a 4-point Likert-type scale, where higher scores indicate greater satisfaction with services received.
Perceived general improvement by the intervention as assessed by the Patient Global Impression of Change scale (PGIC; Guy, 1976) | This single item is only delivered through study completion (approximately 2 months after baseline). Data will be reported once when study is completed (approximately 2 months after baseline)
  Following the IMMPACT (Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials) recommendations, the PGIC will be used to assess the participants' global perceived improvement following treatment. This is a one-item 7-point scale ranging from "very much improved" to "very much worse", with "no change" as the mid-point.
Within-treatment diary | Change in levels of processes at 4 points from baseline through study completion (approximately once every week, prior to each session). Data will be reported once when study is completed (approximately 2 months after baseline)
  At the beginning of each session participants will complete an 8-item diary: 1 item to assess each process of the psychological flexibility hexaflex (willingness, cognitive defusion, contact with present moment, values, committed action and self as context) including an item for pain struggle and pain intensity. Each item is rated on a numerical rating scale of a 1-5 with a specified time-frame (of previous week).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Karekla, Ph.D, Principal Investigator — University of Cyprus

IPD SHARING:
Plan to Share IPD: No